CLINICAL TRIAL: NCT07405450
Title: Clinical Impacts of Structured Robotic Gait Training Programs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Elizabeth Condliffe, PhD MD, Assistant Professor, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: REB22-0511
Record Dates: First submitted 2025-12-12; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Neuromotor Impairments; Walking Impairment
Keywords: Robotic Walking; Trexo

STUDY DESIGN:
Intervention Model Description: All participants will complete robotic walking intervention only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical Impacts of Structured Robotic Gait Training Programs (Experimental): All participants will participate in this arm involving 8 weeks of training 2-3 days/week
  Interventions: Device: Clinical Impacts of Structured Robotic Gait Training Programs

INTERVENTIONS:
Device: Clinical Impacts of Structured Robotic Gait Training Programs — All participants will participate in this arm involving 8 weeks of training 2-3 days/week using the Trexo walking device in clinic

SUMMARY:
Background and Rationale:

Walking impairments impacts the 2-3/1000 children who have cerebral palsy1,2, and others unable to walk due to other central nervous system disorders such as a traumatic brain injury. The impacts of this and related impairment impact all aspects of life. The lifelong costs of these is staggering in terms of dollars (over $1 million/child) and health adjusted life years (~half compared to typically developing populations despite only slightly shorter lifespans). Yet there are currently no effective interventions to treat the fundamental balance impairment that underlie these problems4,5. Early use of robotic gait trainers have shown many benefits6,7, however access to these trainers is limited due to cost, availability, and ease of use within the home. Currently, there are a few options for an overground robotic gait trainer supported by the stability of a walker. The Trexo, is an option designed for use at home or in a community settings, but barriers to access mean that access to this therapy is out of reach for many people who may see benefits.

Research Questions and Objectives:

The aim of this study is to (a) evaluate the feasibility of a clinical robotic gait training program and (b) evaluate the effectiveness of these types of programs in achieving patient, family, and therapist goals. The study will examine adherence to a structured training program to determine if training with a robotic gait trainer in a hospital setting is feasible for the entire length of the designed training program. Goals will be set, a re-evaluation of these goals will be completed following the training program to determine whether or not the clinical program of robotic gait training was successful in helping patients reach the goals set out at the beginning of the program.

DETAILED DESCRIPTION:
Background and Rationale:

Walking impairments impacts the 2-3/1000 children who have cerebral palsy1,2, and others unable to walk due to other central nervous system disorders such as a traumatic brain injury. The impacts of this and related impairment impact all aspects of life. The lifelong costs of these is staggering in terms of dollars (over $1 million/child) and health adjusted life years (~half compared to typically developing populations despite only slightly shorter lifespans). Yet there are currently no effective interventions to treat the fundamental balance impairment that underlie these problems4,5. Early use of robotic gait trainers have shown many benefits6,7, however access to these trainers is limited due to cost, availability, and ease of use within the home. Currently, there are a few options for an overground robotic gait trainer supported by the stability of a walker. The Trexo, is an option designed for use at home or in a community settings, but barriers to access mean that access to this therapy is out of reach for many people who may see benefits.

Research Questions and Objectives:

The aim of this study is to (a) evaluate the feasibility of a clinical robotic gait training program and (b) evaluate the effectiveness of these types of programs in achieving patient, family, and therapist goals. The study will examine adherence to a structured training program to determine if training with a robotic gait trainer in a hospital setting is feasible for the entire length of the designed training program. Goals will be set, a re-evaluation of these goals will be completed following the training program to determine whether or not the clinical program of robotic gait training was successful in helping patients reach the goals set out at the beginning of the program.

Methods:

A prospective, single cohort pragmatic trial to examine the feasibility and utility of Trexo training at Alberta Children's Hospital will be conducted. Participants and their families/caregivers will work with a physiatrist and physiotherapist or kinesiologist with pediatric rehabilitation experience to develop goals and a reasonable training schedule. Clinical training programs will be unique to each participant based on goals and level of function. Consent will be obtained by a member of the research team. Researchers will make it clear that participation in the study is voluntary and that it will not have any effect on their care outside of this program. Participants will be able to provide their own consent if they are 14 years of age or older and have decision making capacity. Parental or guardian consent will be obtained if (i) the participant is 14 years of age or older without decision making capacity or (ii) the participant is younger than 14 years old. We will enroll as many participants into the study as possible within a 2 year time frame. The first visit will be used to determine eligibility, discuss goals, complete a baseline quality of life assessment, and complete an initial fitting. The second visit will be the initial assessment session. The purpose of this visit is to establish a functional baseline for participants before they start training. These will be tailored to each unique participant's goals. After these visits, training will begin. Training visits will be completed as outlined in this clinical program developed by the physiotherapist/kinesiologist. Duration and frequency of the program will depend on goals and feasibility of the training schedule. Following training, the follow-up assessment schedule will repeat the measures taken at the initial assessment session in order to evaluate the success of the training program. Outcome measures will include feasibility of training, usability of the Trexo as a training device, assessment of goals, and adverse events. Feasibility will be assessed by gathering data on therapist training hours, and usability will be assessed via therapist completion of System Usability Scale scoring at two-month intervals during the training period (the open access questionnaire is to be completed via Google Forms questionnaires). Quality of life impact will also be an outcome measure, assessed via the EQ-5D-Y questionnaire (to be administered via a combination of paper forms and electronic Redcap forms). Feasibility outcomes will be presented with descriptive statistics. Assessment of goals will be analyzed using the Wilcoxon signed-rank test for non-parametric difference of means in related samples. The remainder of the analysis plan will focus on descriptive statistics and parameter effect sizes.

ELIGIBILITY:
Inclusion Criteria:

* able to fit into Trexo robotic gait trainer (both leg length and weight); height of <~5'6", weight <150 lbs.)
* able to fulfill training requirements throughout training period
* able to comply with study procedures (assessments, training)
* any age

Exclusion Criteria:

* those with contraindications to training with a robotic gait trainer (ie. medical condition or recent surgery requiring lower extremity immobilization or weight-bearing restriction (ie. fracture, unstable hip subluxation), medical condition requiring a physical activity restriction (ie. unstable arrythmia), pain or symptomatic hypotension while standing, contracture such that the Trexo Robotic Gait Training does not result in forward movement)
* those involved in a potentially confounding intervention (will be discussed case-by-case to determine risk of impacting the study results).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of Sessions Attended | Approximately 8 weeks
  Evaluate the feasibility of using a robotic gait trainer in an out-patient setting by tracking the number of sessions attended by the participants.
Number of Sessions Missed | Approximately 8 weeks
  Evaluate the feasibility of using a robotic gait trainer in an out-patient setting by tracking the number of sessions missed by the participants.
Length of Session | Approximately 8 weeks
  Evaluate the feasibility of using a robotic gait trainer in an out-patient setting by tracking the length of each training session.
Number of steps per session | Approximately 8 weeks
  Evaluate the feasibility of using a robotic gait trainer in an out-patient setting by tracking the number of steps taken by participants in each session.
Clinician time per session | Approximately 8 weeks per participant enrolled.
  Evaluate the feasibility of using a robotic gait trainer in an out-patient setting by tracking the amount of time it takes clinicians to setup, run, and teardown for each training session

SECONDARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | Approximately 8 weeks
  Evaluate the effectiveness of these types of programs in achieving patient, family, and therapist goals, ranked on a 10-point scale (1-10) for performance and satisfaction.
Goal Attainment Scaling (GAS) | Approximately 8 weeks
  Evaluate the effectiveness of these types of programs in achieving patient, family, and therapist goals, ranked on a 5-point scale from -2 to 2 where the midpoint (0) is typically set as baseline and changes are scored based on objectively measured outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
There is an open science plan to share de-identified IPD. All data collected in the study will be de-identified and added to a database. Access by other researchers must be requested and agree to a Terms of Use agreement before access is granted.
Supporting Information: Study Protocol, CSR
Time Frame: Data will become available at the end of the study. There is no plan to close the database.
Access Criteria: Researchers requesting access to the database will be required to sign a Terms of Use agreement.